CLINICAL TRIAL: NCT05421637
Title: Discrepancy Between Perception and Objective Knowledge of Evidence-Based Practice Among Latin American Psychologists: A Cross-Sectional E-Survey Study
Status: Completed | Type: Observational
Sponsor: Universidad Westhill, Facultad de Psicología (Other)
Responsible Party: Principal Investigator, Alejandro Hernández Posadas, Professor of the Faculty of Psychology, University of Americas
Other Study IDs: UW/FP/IC/PSICOLOGIA/2021/003
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Knowledge, Attitudes, Practice; Evidence-based Psychology
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This was a non-experimental, descriptive, prospective and cross-sectional study, for which the CHERRIES checklist was used to report the study in order to improve the quality of the report of such designs. The open-ended survey was voluntary, consisted of 18 items and four sections, the items were not randomized and the survey was estimated to last approximately five minutes.

DETAILED DESCRIPTION:
Sampling:

A non-experimental sampling is carried out by voluntary subjects, since the subjects will come to the study by a call for applications.

Sample size

The formula of infinite population of qualitative variables will be used, because we will work with ordinal variables and because the total number of observation units that integrate it is unknown or when its population is greater than 100,000 and the formula is the following:

The sample size for 100,000 people should be 384 people, so that 95% of the time the data you want to measure is in the interval ±5% with respect to the data observed in the evaluation.

Data management plan:

Data dictionary design

Training will be provided and data dictionary will be developed describing the properties of variables such as data type (e.g. string and number), variable size, data encoding, and constraints and validations attached to a given variable (Annex).

Data collection

The research data will be obtained through the Google forms, which has "SOC 2" accreditation that meet best practices and security, as they are transmitted over a secure HTTPS connection and that user logins were protected through TLS. Furthermore, data is encrypted using industry and research standard encryption algorithms.

Data Retention

The database will be generated in Excel for further analysis in R studio, which will be kept at the University on an encrypted USB stick for data security and the password to this stick will only be held by the project manager.

Standards that provide data integrity, accuracy and coherence

The International Classification of Diseases (ICD- 11) will be used to present data consistency, accuracy and completeness through the optimal definition of mental health entities. On the other hand, the standards for data use recommended by The Global Health Training Centre will be used:

(a) The column heading (variable) is not changed between data. b) The same terminology is maintained for all variables. c) There is a consistent format and standard definition for subject identification.

d) The name of the datasets is always the same. e) Name of the form / CRF section, e.g., demographic data f) A list of data objects (names and definitions) g) Description of the data element in natural language h) Detailed properties of the data elements (data type, size, nullability, optionality, indexes) i) Response options, e.g., check box, radio button, text j) Validation rule(s), e.g., required field, range checking k) Relationship of data elements to other data elements. l) Details about the privacy and security restrictions that should be associated with the element, e.g., Protected Health Information status.

Methodological guidelines for reporting the study:

The guide to improve the quality of methodological reporting of cross-sectional online studies called CHERRIE will be used.

Data analysis

Descriptive statistics were used to analyze the central tendency frequencies of the participants' characteristics. Non-parametric analyses will be applied because the data do not meet the criteria of normality in the analysis of their distribution, the type of variable and the number of participants; therefore, Spearman correlations will be used to contrast ordinal data. On the other hand, we plan to use odds ratio analysis to determine the possibility that knowledge of evidence-based psychology is present in one population group with more studies than in another.

ELIGIBILITY:
Inclusion Criteria:

* Be an active psychology student at any university in Latin America.
* To have completed at least one semester of the psychology degree program
* Be between 18 and 65 years of age
* Be able to read and write
* Be a native Spanish speaker
* Agree to participate voluntarily in the study.
* Sign the informed consent form

Exclusion Criteria:

* Not currently residing in any Latin American country.
* Those persons who have not studied psychology and are performing related activities.
* Repeated IP (Internet Protocol)
* Marginal frequencies in the sociodemographic data.
* Participants who do not answer the complete scales.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Latin American psychologists of all specialties and degrees of studies.
Sampling Method: Non-Probability Sample
Enrollment: 1506 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Knowledge of evidence-based PSychology | 1 month
  To explore knowledge in evidence-based psychology, the studies conducted by the American Psychological Association (2005) and the studies conducted by Gaxiola-Pérez et al. (2019) were used as a basis, so that the components, phases that compose it, tools for critical reading and levels of evidence were questioned, in order to create a questionnaire of four items for the evaluation of knowledge, where the maximum score was four and the minimum value was zero.
Perception of Evidence-based Psychology | 1 month
  The perception was assessed using a visual analog scale, according to the methodological recommendations for instruments that assess online perception and considered: a) Degree of familiarity, b) Importance attached to it, and c) Frequency with which it is applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Westhill University, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No